CLINICAL TRIAL: NCT05895240
Title: MUNI-SEP TRIAL-The Role of Ulinastatin in Preventing Severe Sepsis and Consequent Morbidities and Mortality; A Randomized Clinical Trial in Pakistan.
Brief Title: Role of Ulinastatin in Preventing Severe Sepsis and Consequent Morbidities and Mortality
Acronym: MUNI-SEP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, ZA, Associate Professor, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NO.F.2-81/2022-GENL/229/JPMC
Record Dates: First submitted 2023-05-13; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Severe Sepsis; Septic Shock; MODS
MeSH Terms: conditions — Sepsis; Shock, Septic; Multiple Organ Failure | interventions — urinastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group Arm (No Intervention): Standard of care treatment arm, study medication will not be given
- Active Intervention Arm (Experimental): This group will receive Nine MiU Ulinastatin in three divided doses 8 hourly
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin — Nine MiU Ulinastatin in three divided doses 8 hourly for 3-5 days
  Arms: Active Intervention Arm

SUMMARY:
The study will enhance the theory in the frame of reference on the efficacy of Ulinastatin while managing sepsis and subsequent morbidity and mortality. Moreover, the present study will explore Ulinastatin's prophylactic role in progression of multiple organ dysfunctions. Furthermore, the study will have the clinical implications in predicting the ICU admitted patient's stay and related cost in the context of new drug. Current researches will explore the new dimensions in Pakistan's healthcare facilities, paving the way of future academics to analyze it in order to enhance healthcare outcomes.

DETAILED DESCRIPTION:
The current study is a randomised clinical trial with the aim of exploring the following objectives in the context of Pakistan:

* To determine the efficacy of Ulinastatin in preventing the progression of Sepsis to Severe Sepsis and septic shock.
* To assess the role of Ulinastatin in preventing the onset of MODS in sepsis-induced patients.
* To investigate the impact of Ulinastatin on sepsis associated mortality and morbidity.
* To explore the role of Ulinastatin in reducing ICU stays and associated costs in defined patients.
* To provides a condensed basis to understand ULINASTATIN as a sepsis management drug.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 or <60
* Sepsis, and severe sepsis, as defined in operational definitions
* Patients voluntarily agreed to participate in the study after informed consent

Exclusion Criteria:

* Fulminant hepatic failure
* Acute cerebrovascular accidents
* Acute poisoning
* Chronic Kidney Disease stage 5
* Diagnosed case of immune thrombocytopenia
* Low output cardiac failure, with left ventricular ejection fraction <20%
* Advance chronic obstructive pulmonary disease on long term oxygen therapy
* Lactation or pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Prevention of MOD's in patients with sepsis | Day 1 of enrollment
  To assess the role of Ulinastatin in preventing the onset of MODS in sepsis-induced patients. Sepsis is defnied as evidence of infection (positive culture of blood, Urine, Tracheal) or suspected infection (by a physician) plus 2 out of 4 criteria's of SIRS. MODS is presence of two or more organ dysfunction with scoring ≥2 of each organ as per Sequential Organ Failure Assessment (SOFA) score.
Prevention of MOD's in patients with sepsis | Day 3 of enrollment
  To assess the role of Ulinastatin in preventing the onset of MODS in sepsis-induced patients. Sepsis is defnied as evidence of infection (positive culture of blood, Urine, Tracheal) or suspected infection (by a physician) plus 2 out of 4 criteria's of SIRS. MODS is presence of two or more organ dysfunction with scoring ≥2 of each organ as per Sequential Organ Failure Assessment (SOFA) score.
Prevention of MOD's in patients with sepsis | Day 5 of enrollment
  To assess the role of Ulinastatin in preventing the onset of MODS in sepsis-induced patients. Sepsis is defnied as evidence of infection (positive culture of blood, Urine, Tracheal) or suspected infection (by a physician) plus 2 out of 4 criteria's of SIRS. MODS is presence of two or more organ dysfunction with scoring ≥2 of each organ as per Sequential Organ Failure Assessment (SOFA) score.
Effect on in-hospital mortality | During first 48 hours of hospital stay after enrollment
  To investigate the impact of Ulinastatin on sepsis associated mortality.
Effect on 7 days mortality | During the 7 days of enrollment
  To investigate the impact of Ulinastatin on sepsis associated mortality.
Effect on 14 days mortality | During the 14 days of enrollment
  To investigate the impact of Ulinastatin on sepsis associated mortality.
Effect on 28 days mortality | During the 28 days of enrollment
  To investigate the impact of Ulinastatin on sepsis associated mortality.

SECONDARY OUTCOMES:
Number of days on mechanical ventilation | Up to 28 days after enrollment
  To explore the role of Ulinastatin in reducing the number of days on mechanical ventilation
Number of days in ICU | Up to 28 days after enrollment
  To explore the role of Ulinastatin in reducing ICU stays.
Prevention of Severe Sepsis in patients admitted with Sepsis | Up to 28 days after enrollment
  To determine the efficacy of Ulinastatin in preventing the progression of sepsis to severe sepsis. Severe sepsis is sepsis as defined above plus at least one organ/system dysfunction scoring ≥ 2 as per Sequential Organ Failure Assessment (SOFA) score.
Prevention of Septic Shock in patients admitted with Sepsis | Up to 28 days after enrollment
  To determine the efficacy of Ulinastatin in preventing the progression of sepsis to septic shock. Septic shock is persistent hypotension requiring vasopressors to maintain mean arterial pressure of 65mmHg or higher and a serum lactate level greater than 2mmol/L despite adequate volume resuscitation with 30ml/kg of crystalloid solution.

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Ali, FCPS, Principal Investigator — Jinnah Postgraduate Medical Centre Karachi
Locations (1):
- Medical ICU, Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No